CLINICAL TRIAL: NCT07188142
Title: Investigating the Effects of Two Different Desensitizing Agents on Mitigating Post-Operative Sensitivity Following Composite Restorations - a Randomized Controlled Trial
Brief Title: Gluma Compared With Bonding Agent for Post-operative Sensitivity Following Composite Restorations
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beenish Hassan (Other)
Responsible Party: Sponsor-Investigator, Beenish Hassan, Post Graduate Trainee, Margalla Institute of Health Sciences
Organization: Margalla Institute of Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DB/272/25
Record Dates: First submitted 2025-09-13; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Post-operative Sensitivity; Dentin Hypersensitivity; Dental Caries; Tooth Sensitivity After Composite Restorations; Post-operative Sensitivity After Class I Composite Restorations
Keywords: Post-operative sensitivity; Dentinal hypersensitivity; Class I caries; Gluma desensitizer; Composite restoration
MeSH Terms: conditions — Dentin Sensitivity; Dental Caries | interventions — Gluma; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Comparator: Group A (Gluma Desensitizer Group) (Active Comparator): Patients receiving Gluma desensitizer followed by universal bonding agent and composite restoration on Class I carious lesions.
  Interventions: Drug: Drug/Agent: Gluma Desensitizer
- Active Comparator: Group B (Control Group) (Active Comparator): Patients receiving universal bonding agent and composite restoration without Gluma desensitizer on Class I carious lesions.
  Interventions: Drug: Drug/Agent: No desensitizer (Control)

INTERVENTIONS:
Drug: Drug/Agent: Gluma Desensitizer — Gluma desensitizer applied to prepared tooth surface, followed by universal bonding agent and composite restoration. Application done during the first visit of restorative treatment. Post-operative sensitivity measured at baseline, 1 week, 1 month, and 3 months.
  Other Names: Gluma; Glutaraldehyde/HEMA solution; Dentin desensitizer
  Arms: Active Comparator: Group A (Gluma Desensitizer Group)
Drug: Drug/Agent: No desensitizer (Control) — Universal bonding agent applied followed by composite restoration without prior use of Gluma desensitizer. Post-operative sensitivity measured at baseline, 1 week, 1 month, and 3 months.
  Other Names: Control group; Composite restoration without desensitizer
  Arms: Active Comparator: Group B (Control Group)

SUMMARY:
* The aim of this study is to compare the effectiveness of Gluma desensitizer in reducing post-operative sensitivity following composite restorations in posterior teeth. -Patients visiting OPD will be selected after fulfilment of inclusion criteria. Patients aged 18-45 meeting inclusion criteria and presenting with active primary class I carious lesions on vital molar teeth with ICDAS score 3 will be randomly assigned into two groups: -Group A: Patients will be provided with Gluma desensitizer, Universal Bonding agent and Composite restoration and -Group B: Patients will receive Universal bonding agent and Composite restoration. -The progress of treatment will be followed up immediately (baseline) and at regular follow up visits at 1 week, 1 month and 3 months.
* Post-operative sensitivity will be assessed using an air stimulus and rated on a numeric rating scale for post-operative sensitivity assessment ranging from 0 to 10.

DETAILED DESCRIPTION:
-This randomized clinical trial is done to compare the effectiveness of Gluma desensitizer in reducing post-operative sensitivity following composite restorations in posterior teeth. -The study sample size includes a total of 60 participants aged 18 to 45, each having two Class I carious lesions requiring composite restorations. -Patients will be randomly divided into two groups using a lottery method: -Group A receiving Gluma desensitizer, universal bonding agent, and composite restoration, and -Group B receiving universal bonding agent and composite restoration without desensitizer. -Patients will be selected from the outpatient dental clinic after fulfilling inclusion criteria, which include age between 18 and 45 years, good oral hygiene, active primary Class I carious lesions on vital molar teeth with an ICDAS score of 3, complaints of sensitivity to air and osmotic stimulus, positive response to cold test, and no signs of pulp inflammation or spontaneous pain before treatment. -Exclusion criteria include excessive tooth wear due to clenching or abnormal habits, traumatic occlusion, periodontal or gingival disease, and current use of analgesics and/or anti-inflammatory medication. -Post-operative sensitivity will be measured clinically using an air stimulus and evaluated on a numeric rating scale for post-operative sensitivity assessment ranging from 0 to 10. ranging from 0 (no sensitivity) to 10 (unbearable sensitivity) at baseline (immediately after treatment) and at 1 week, 1 month, and 3 months postoperatively. -Statistical analysis will be performed using non-parametric tests including the Friedman test for within-group comparisons and Wilcoxon signed-rank test for between-group differences, with significance set at p < 0.05. -This study will further add to the literature by providing clinical evidence regarding the efficacy of Gluma desensitizer in reducing post-operative sensitivity and improving patient comfort following restorative dental procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-45 years.
* Good oral hygiene.
* Active primary class I carious lesions on vital molar teeth with ICDAS score 3
* Patients complaining of sensitivity to air and osmotic stimulus.
* Teeth having a positive cold test.
* No signs of pulp inflammation or spontaneous pain before treatment.

Exclusion Criteria:

* Excessive tooth wear due to clenching or abnormal habits.
* Traumatic occlusion.
* Periodontal or gingival disease.
* Patients using analgesics and/or anti-inflammatory medicine.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative sensitivity | 3 months
  Change in dentinal hypersensitivity following Class I composite restorations, measured using a numeric rating scale to evaluate Post-operative Sensitivity (0-10) (0: No sensitivity, 10: Unbearable sensitivity) in response to air stimulus at baseline, 1 week, 1 month and 3 months post-treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Margalla Institute of Health Sciences Quaid e Azam Avenue, Gulraiz phase 3, Gulraiz Housing Scheme, Rawalpindi, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No